CLINICAL TRIAL: NCT05867875
Title: Impact of the Non-invasive Oxygen-reserve-index (ORI) Versus Standard of Care on Peripheral Oxygen Saturation (SpO2) During Endotracheal Intubation (ETI) in Intensive Care Unit: Randomised Superiority Multi-center 2 Arms, Open Trial
Brief Title: Non-invasive Early Oxygen- Reserve-index (ORI) Determination to Prevent Hypoxaemia During Endotracheal Intubation
Acronym: NESOI-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RC22_0506
Record Dates: First submitted 2023-04-27; First posted 2023-05-22 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Intensive Care Unit
Keywords: ORI; intensive care unit; ETI; Masimo Rad7

STUDY DESIGN:
Intervention Model Description: Consecutive Intensive Care Unit (ICU) patients requiring ETI will be randomly allocated to ETI with or without ORI monitoring before beginning of preoxygenation, with stratification by centre, expert or nonexpert intubator status (experts: ≥5 years' ICU experience, or ≥1 year ICU experience plus ≥2 years' anaesthesiology training), and Non-Invasive Ventilation (NIV) or others devices for preoxygenation. Randomisation will be via an electronic case-report form, using a balanced scheme with stratification as described above.
Who Masked: Investigator
Masking Description: During intubation procedure, blinded continuous monitoring of SpO2 and ORI (for control group) will be performed by appropriate monitor (Masimo Rad7) with data extraction at regular intervals.
  Oxygen saturation will be tracked during ETI by research nurse or assistant nurse dedicated to fill the eCRF. ORI evolution will not be provided to investigators in the standard of care group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (ORI) (Experimental): ORI and SpO2 monitoring values during preoxygenation of patients will be provided to investigator to determine anaesthesia induction initiation. Anesthesic induction is provided after 30 secondes at ORI > 0.6 and at least 2 min 30 of preoxygenation (so globaly 3 minutes of preoxygenation)
  Interventions: Other: Unblinded ORI values
- Standard of care (SoC) group (Other): Only SpO2 values during preoxygenation of patients will be provided to investigator to determine anaesthesia induction initiation. Anesthesic induction is provided at least 3 min of preoxygenation
  Interventions: Other: Blinded ORI values

INTERVENTIONS:
Other: Unblinded ORI values — ORI and SpO2 monitoring will be performed using Masimo Rad 7 and both values will be provided to investigator
  Arms: Experimental group (ORI)
Other: Blinded ORI values — ORI and SpO2 monitoring will be performed using Masimo Rad 7 and only SpO2 values will be provided to investigator
  Arms: Standard of care (SoC) group

SUMMARY:
The purpose of this study is to determine whether ORI monitoring increases the lowest oxygen saturation level during the interval between the first laryngoscopy (defined as introduction of the laryngoscope into the mouth) and the end of the second minute after successful ETI.

DETAILED DESCRIPTION:
The trial population will be adults (18 years of age or older) who need endotracheal intubation while hospitalized in ICU

ELIGIBILITY:
Inclusion Criteria:

* ICU admission and need for ETI to allow mechanical ventilation
* Need for supplemental oxygen (via any device and at any flow rate) to obtain SpO2>97%
* Patient or next of kin informed about the study and having consented to participation of the patient in the study (patients with coma are unable to consent). If patient is no competent and no next of kin can be contacted during screening for the study, trial inclusion will be completed as an emergency procedure by the ICU physician, in compliance with French law
* Patients affiliated to a social security system

Exclusion Criteria:

* Patients participating in intubation research with an oxygenation endpoint will not be eligible for inclusion
* Fiberoptic intubation required according to physician in charge
* Contra-indications to laryngoscopy (e.g., unstable spinal lesion)
* Insufficient time to include and randomise the patient (e.g., because of cardiac arrest)
* Age <18 years
* Currently pregnant or breastfeeding
* Correctional facility inmate
* Under guardianship, curatorship or under protection of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 950 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-05-26 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Determine whether ORI monitoring increases the lowest oxygen saturation level during ETI | From the first laryngoscopy (defined as introduction of the laryngoscope into the mouth) until the end of the second minute after successful ETI
  Lowest oxygen saturation is monitored by Masimo Rad7 oximeter during ETI in Experimental and Control groups

SECONDARY OUTCOMES:
Determine whether ORI monitoring increases the lowest oxygen saturation level according to local oximeter. | From the first laryngoscopy (defined as introduction of the laryngoscope into the mouth) until the end of the second minute after successful ETI
  Lowest oxygen saturation monitored by local oximeter during ETI in Experimental and Control groups are compared to values monitored by Masimo Rad7 in same conditions
Determine whether ORI monitoring increases the lowest oxygen saturation level during ETI in "Body Mass Index (<30 or ≥30)" subgroup | From the first laryngoscopy (defined as introduction of the laryngoscope into the mouth) until the end of the second minute after successful ETI
  Lowest oxygen saturation is monitored by Masimo Rad7 oximeter during ETI in "Body Mass Index" subgroup

OTHER OUTCOMES:
Determine whether ORI monitoring increases the lowest oxygen saturation level during ETI in "Reason for ETI (hypoxaemia/other)" subgroup | From the first laryngoscopy (defined as introduction of the laryngoscope into the mouth) until the end of the second minute after successful ETI
  Lowest oxygen saturation is monitored by Masimo Rad7 oximeter during ETI in "Reason for ETI (hypoxaemia/other)" subgroup
Determine whether ORI monitoring increases the lowest oxygen saturation level during ETI in "Shock/No shock (at inclusion)" subgroup | From the first laryngoscopy (defined as introduction of the laryngoscope into the mouth) until the end of the second minute after successful ETI
  Lowest oxygen saturation is monitored by Masimo Rad7 oximeter during ETI in "Shock/No shock (at inclusion)" subgroup
Determine whether ORI monitoring increases the lowest oxygen saturation level during ETI in "Difficult Intubation (yes or no)" subgroup | From the first laryngoscopy (defined as introduction of the laryngoscope into the mouth) until the end of the second minute after successful ETI
  Lowest oxygen saturation is monitored by Masimo Rad7 oximeter during ETI in "Difficult Intubation (yes or no)" subgroup
Determine whether ORI monitoring increases the lowest oxygen saturation level during ETI in "ORI threshold (<0.6 or ≥0.6)" subgroup | From the first laryngoscopy (defined as introduction of the laryngoscope into the mouth) until the end of the second minute after successful ETI
  Lowest oxygen saturation is monitored by Masimo Rad7 oximeter during ETI in "ORI threshold (<0.6 or ≥0.6)" subgroup
Assess safety of ORI monitoring | From the first laryngoscopy (defined as introduction of the laryngoscope into the mouth) until the end of the second minute after successful ETI
  Occurrence of at least one severe life-threatening complication (death, cardiac arrest, arterial systolic pressure <90 mmHg, and/or SpO2<80%) and occurrence of each are assessed in Experimental and Control group
Assess efficacy of ORI monitoring on ICU mortality | From the first laryngoscopy (defined as introduction of the laryngoscope into the mouth) until discharge from intensive care unit or up to 28 days
  ICU mortality is assessed in Experimental and Control groups
Assess efficacy of ORI monitoring on 28-day mortality | From the first laryngoscopy (defined as introduction of the laryngoscope into the mouth) until day 28
  28-day mortality is assessed in Experimental and Control groups
Assess efficacy of ORI monitoring on ICU stay length | From the first laryngoscopy (defined as introduction of the laryngoscope into the mouth) until discharge from intensive care unit or up to 28 days
  ICU stay length is assessed in Experimental and Control groups
Assess efficacy of ORI monitoring on hospital stay length | From the first laryngoscopy (defined as introduction of the laryngoscope into the mouth) until discharge from hospital or up to 28 days
  Hospital stay length is assessed in Experimental and Control groups
Assess efficacy of ORI monitoring on Mean Cognitive Core at day 28 (modified Telephone Interview for Cognitive Status) | Day 28
  Mean Cognitive Score at day 28 using modified Telephone Interview for Cognitive Status is assessed in Experimental and Control groups Values range from 0 to 43, with higher scores indicating better cognition

CONTACTS AND LOCATIONS:
Locations (21):
- France (21):
  - CHU Angers, Angers
  - CH Argenteuil, Argenteuil
  - CHU Bordeaux, Bordeaux
  - CH du Cotentin, Cherbourg
  - CH Cholet, Cholet
  - APHP - Hôpital Louis Mourier, Colombes
  - CHU de Dijon, Dijon
  - CH d'Haguenau, Haguenau
  - CHD Vendée, La Roche-sur-Yon
  - CH de Versailles, Le Chesnay
  - CHR Lille - Hôpital Roger Salengro, Lille
  - HCL - Hôpital Edouard Herriot, Lyon
  - CHU de Nantes, Nantes
  - CHU de Nice, Nice
  - CHR d'Orléans, Orléans
  - Hôpital Saint-Louis, Paris
  - APHP - Hôpital Cochin, Paris
  - CHU de Rennes, Rennes
  - CH de Roanne, Roanne
  - CHRU de Strasbourg, Strasbourg
  - CHRU de Tours, Tours

REFERENCES:
- [Derived] Hille H, Le Thuaut A, Asfar P, Quelven Q, Mercier E, Le Meur A, Quenot JP, Lemiale V, Muller G, Cour M, Ferre A, Berge A, Curtiaud A, Touron M, Plantefeve G, Chakarian JC, Ricard JD, Colin G, Orieux A, Girardie P, Jozwiak M, Rouaud M, Juhel C, Reignier J, Lascarrou JB; CRICS-TRIGGERSEP Network. Impact of non-invasive oxygen reserve index versus standard SpO2 monitoring on peripheral oxygen saturation during endotracheal intubation in the intensive care unit: Protocol for the randomized controlled trial NESOI2. PLoS One. 2024 Sep 16;19(9):e0307723. doi: 10.1371/journal.pone.0307723. eCollection 2024. PMID 39283873